CLINICAL TRIAL: NCT03391401
Title: Investigation of Microbiome-based Prognostical Biomarkers in Patients With Morbid Obesity and Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Collaborators: University of Bonn (Other)
Responsible Party: Principal Investigator, Andreas Plamper, Assistant study director, St. Franziskus Hospital
Other Study IDs: 2017110
Record Dates: First submitted 2017-12-07; First posted 2018-01-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; NAFLD; Microbiome
MeSH Terms: conditions — Obesity, Morbid; Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hair samples, blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adip1: Patients with morbid obesity (i.e. BMI >35 kg/sqm) and age >18 scheduled for bariatric surgery (all standard procedures included)
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Any bariatric operation that is considered as a standard procedure in bariatric surgery (i.e. sleeve gastrectomy, roux-en-y gastric bypass, mini-gastric / one anastomosis gastric bypass, redo and revisional bariatric surgery).

SUMMARY:
Morbid obesity leads to non-alcoholic fatty liver disease (NAFLD), and not all NAFLD cases benefit from weight loss e.g. after bariatric surgery. Our aim is to find out, which intrahepatic factors and / or biomarkers might be beneficial or can be identified as prognostic factors for remission of NAFLD after weight loss. As other factors such as the microbiome or muscle and fatty tissue also influence the development of obesity and liver diseases, it is planned to examine these parameters before and after bariatric surgery as well.

Tissue biopsies will therefore be taken during the surgery, and blood as well as stool samples will be collected and compared for suitable biomarkers before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 40 kg/sqm or
* BMI above 35 kg/sqm and comorbidities related to morbid obesity (e.g. type 2 diabetes, hypertension, coronary heart disease, dyslipoproteinemia, sleep apnea, and others

Exclusion Criteria:

* BMI below 35 kg/sqm
* no informed consent
* patient not suitable for bariatric surgery (severe psychological disorder, pregnancy, drug abuse, active malignant or other consuming disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients with the above given criteria that are willing to treat their morbid obesity by bariatric surgery and have at least absolved 3 months of failed conservative treatment for morbid obesity, have shown to have good long-time compliance and high motivation.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Changes of microbiome after bariatric surgery | at time of operation, 3 and 6 months after the operation
  Collection of stool sample before and after (3 and 6 months) the operation
Changes of microbiome after bariatric surgery | at time of operation, 3 and 6 months after the operation
  Collection of blood sample before and after (3 and 6 months) the operation

SECONDARY OUTCOMES:
incidence of fatty liver in obese patients | during the operation
  Surgical liver biopsy during laparoscopy

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University of Bonn, Bonn
  - St. Franziskus-Hospital, Cologne

REFERENCES:
- [Result] Li Z, Bowerman S, Heber D. Health ramifications of the obesity epidemic. Surg Clin North Am. 2005 Aug;85(4):681-701, v. doi: 10.1016/j.suc.2005.04.006. PMID 16061080
- [Result] Reeves GK, Pirie K, Beral V, Green J, Spencer E, Bull D; Million Women Study Collaboration. Cancer incidence and mortality in relation to body mass index in the Million Women Study: cohort study. BMJ. 2007 Dec 1;335(7630):1134. doi: 10.1136/bmj.39367.495995.AE. Epub 2007 Nov 6. PMID 17986716
- [Result] Sjostrom L, Peltonen M, Jacobson P, Sjostrom CD, Karason K, Wedel H, Ahlin S, Anveden A, Bengtsson C, Bergmark G, Bouchard C, Carlsson B, Dahlgren S, Karlsson J, Lindroos AK, Lonroth H, Narbro K, Naslund I, Olbers T, Svensson PA, Carlsson LM. Bariatric surgery and long-term cardiovascular events. JAMA. 2012 Jan 4;307(1):56-65. doi: 10.1001/jama.2011.1914. PMID 22215166
- [Result] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Result] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Result] Henao-Mejia J, Elinav E, Jin C, Hao L, Mehal WZ, Strowig T, Thaiss CA, Kau AL, Eisenbarth SC, Jurczak MJ, Camporez JP, Shulman GI, Gordon JI, Hoffman HM, Flavell RA. Inflammasome-mediated dysbiosis regulates progression of NAFLD and obesity. Nature. 2012 Feb 1;482(7384):179-85. doi: 10.1038/nature10809. PMID 22297845
- [Result] Fujisaka S, Ussar S, Clish C, Devkota S, Dreyfuss JM, Sakaguchi M, Soto M, Konishi M, Softic S, Altindis E, Li N, Gerber G, Bry L, Kahn CR. Antibiotic effects on gut microbiota and metabolism are host dependent. J Clin Invest. 2016 Dec 1;126(12):4430-4443. doi: 10.1172/JCI86674. Epub 2016 Oct 24. PMID 27775551
- [Result] Mathis D. Immunological goings-on in visceral adipose tissue. Cell Metab. 2013 Jun 4;17(6):851-859. doi: 10.1016/j.cmet.2013.05.008. PMID 23747244